CLINICAL TRIAL: NCT00424736
Title: Role of Whole Body Imaging in Asymptomatic Pediatric Trauma Patients
Brief Title: the Role of Total Body Imaging in Asymptomatic Pediatric Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: igorjer1
Record Dates: First submitted 2007-01-16; First posted 2007-01-19 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Injuries and Wounds
Keywords: blunt trauma, pediatric patient, imaging, computer tomography
MeSH Terms: conditions — Wounds and Injuries; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: whole body CT scan

SUMMARY:
Whole body imaging has no role in asymptomatic pediatric trauma patients

DETAILED DESCRIPTION:
Negative physical examination alone has been shown unreliable for excluding intra-abdominal injuries in adult patients with multitrauma. Therefore, the management of patients with a normal clinical examination after blunt trauma is a subject of controversy. Since 1970s, computer tomography (CT) has become the mainstay of evaluating hemodynamically stable trauma patients. It's generally accepted that hemodynamically stable patient with abnormal abdominal examination results require the use of CT as well as patients with depressed level of consciousness. Controversy exists with the awake, clinically evaluable patients with no obvious signs of abdominal and chest trauma. In the last years number of studies express CT role in evaluation of asymptomatic trauma patient with mechanism of injury supporting probability of internal organs injury. Those studies show that in a large number of patients the management was changed according to CT results. The authors recommended liberal use of CT in trauma patient population. All those studies have been performed in adult trauma patients. The purpose of this study is to evaluate the role of whole body imaging in pediatric patients with suspicious mechanism of injury, which are hemodynamically stable and has no obvious signs of chest and abdominal injury. The incidence of injury in these patient population as well as changes in treatment based on results of CT will be examined. Methods The prospective observational study will be performed in Assaf Harofeh Medical Center. All patients up to 15 years old with blunt mechanism of multisystem trauma will be eligible for enrollment to the study. Only patients whose parents singed the inform consent will be enrolled.Inclusion criteria will be based on the mechanism of injury: 1. no visible injury of chest and abdomen2. hemodynamically stable3. normal abdominal examination in neurologically intact patient or unevaluable abdominal examination in patients with depressed level of consciousness. 4. significant mechanism of injury as any of the following a. high speed (more than 55km/hr) motor vehicle accident b. fall of greater than 3 meters c. automobile hitting pedestrian d. assaulted with depressed level of consciousness All patients will undergo CT of the head, chest, abdomen and pelvis as a part of their evaluation. CT scan will be performed in Emergency Department short after patient's admission and clinical evaluation. An abnormal CT will be defined as exhibiting any traumatic abnormality. Patient treatment plan changes will be defined as alteration in management based directly on CT findings.Data regarding patient demographics, mechanism of injury, physical examination findings, Glasgow Coma Score on emergency department admission, Injury Severity Score, radiologic interpretation of chest and pelvic roentgenograms, injuries required operative procedures, laboratory data, CT scan findings, and changes in management plan based on CT findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All asymptomatic trauma patients from 0 to 15 years old

Exclusion Criteria:

* Any pediatric trauma patients with clinical indications for CT scan

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Igor Jeroukhimov, MD, Principal Investigator — Assaf-Harofeh Medical Center